CLINICAL TRIAL: NCT00423215
Title: An Open Therapeutic Observational Evaluation of the Efficacy and Safety Profile of Lantus in Everyday Medical Practice in Type 2 Diabetes Mellitus Patients, Who Start Receiving Lantus - Treated With Any Other Insulin, With A1c>7%
Brief Title: LAPAS Study: Insulin Glargine in Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Other Study IDs: HOE901_5062
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2009-06-15 (Estimated); Status verified 2009-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Type II diabetes
  Interventions: Drug: Insulin glargine (LANTUS)

INTERVENTIONS:
Drug: Insulin glargine (LANTUS) — The patients will receive Lantus administered by subcutaneous injection, once daily at any time but at the same time each day.
  Treatment duration: 4 months.

SUMMARY:
The objective of this protocol is to confirm the efficacy and safety profile of Lantus in every day medical practice, in type 2 diabetic patients, have been treated with any other insulin but who did not reach the target of A1c = 7%.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus,
* Having been treated with any other insulin, but who did not reach the target of A1c=7%.
* Ability and willingness to perform Self Monitoring Blood Glucose measurement

Exclusion Criteria:

* Will follow the prescribing information (Summary of Product Characteristics).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Type II Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 1007 (Actual)
Dates: Start 2006-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Measure of Glycolysated Haemoglobin (HbA1c) level reduction | Delta between the treatment start and the end of the study (i.e. 4 months +/- 2 weeks)

SECONDARY OUTCOMES:
Measure of Fasting Blood Glucose (FBG) level reduction | Delta between the treatment start and the end of the study (i.e. 4 months +/- 2 weeks)
Investigator assessment | At the end of the study (i.e. 4 months +/- 2 weeks)
Insulin dose | At the end of the study (i.e. 4 months +/- 2 weeks)
Patient's satisfaction | At the end of the study (i.e. 4 months +/- 2 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Nurit Tweezer-Zaks, M.D., Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Netanya, Israel